CLINICAL TRIAL: NCT04226872
Title: Supporting Family Caregivers of Persons Living With Dementia: Effectiveness and Sustainability of My Tools 4 Care-In Care
Brief Title: Supporting Family Caregivers of Persons Living With Dementia: Effectiveness and Sustainability of MT4C-In Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00090771
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-09

CONDITIONS: Dementia; Family
Keywords: Caregivers; Quality of life; Dementia; Web-based intervention
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive access to My Tools for Care - In Care for 2 months. They will also receive a copy of the Alzheimer Society's "The Progression Of Alzheimer's Disease - Overview Booklet".
  Interventions: Behavioral: My Tools for Care - In Care
- Control (No Intervention): The control group will not receive the intervention (i.e. they will not access My Tools for Care - In Care). They will receive a copy of the Alzheimer Society's "The Progression Of Alzheimer's Disease - Overview Booklet". Data collection for outcome variables will be the same as participants in the intervention group.

INTERVENTIONS:
Behavioral: My Tools for Care - In Care — Self-administered web-based transition toolkit (My tools 4 Care - In Care) contains interactive activities and resources to help carers through transitions that they face after the person living with dementia has moved to a long-term care setting.
  Arms: Intervention

SUMMARY:
When a person living with dementia moves into a long term care facility, their family members remain involved in their care. They learn new roles and make significant and often stressful adjustments. These caregivers are an at-risk group, and evidence suggests that their mental health may actually worsen after the person they are caring for moves into long term care. The research team previously created a free, web-based, interactive, intervention called My Tools 4 Care-In Care (MT4C-In Care) and tested it with 37 caregivers in Alberta. Caregivers found the toolkit to be easy to use, feasible, acceptable, and satisfactory, and reported increased hope and decreased loss and grief, after using it. Additionally, they reported that the toolkit helped them through the transitions they experience when their family member lives in long term care.

In this next study we want to see if MT4C-In Care can improve the quality of life, hope, social support, self-efficacy, and decrease the loss, grief and loneliness of family caregivers. During phase 1 the existing MT4C-In Care toolkit was reviewed with input from family caregivers of persons living with dementia in long term care through focus group interviews. The toolkit is now being revised and will be tested, during phase 2, with 280 caregivers of persons living with dementia in long term care across 4 provinces in Canada (Alberta, Ontario, Saskatchewan, and Manitoba). These caregivers will be randomly assigned into an intervention (caregivers with access to MT4C-In Care) and a control group (no access to MT4C-In Care).

DETAILED DESCRIPTION:
Background: Caregivers of Persons Living with Dementia (PLWD) in a Long Term Care (LTC) community are an at-risk group, and evidence suggests that the caregiver's mental health may actually worsen after the PLWD moves to LTC. Caregivers may report feelings of blame, self-doubt, loneliness, isolation, and powerlessness which negatively affect their mental health. This at-risk group requires support to maintain and improve their quality of life. My Tools 4 Care - In Care (MT4C-In Care) is a self-administered, multicomponent, flexible, and interactive website designed specifically to support family caregivers of PLWD in LTC to address this gap in service and the significant concerns about their mental health. The feasibility study in Alberta demonstrated that MT4C-In Care is informative, convenient, and easy to use; and shows potential to help caregivers cope with the transitions and adjustments beyond the PLWD's admission to LTC, increasing caregivers' hope and decreasing their loss and grief.

Purpose: The purpose of Phase 2 is to implement and evaluate MT4C-In Care to assess its effectiveness, and the influence of participant factors (i.e., gender, cultural background, age, etc.) on the use of MT4C-In Care across four Canadian provinces (Alberta, Saskatchewan, Manitoba, and Ontario). The ability of MT4C-In Care to improve hope, self-efficacy, quality of life, social support, and mental health, and decrease grief and loneliness will be rigorously assessed in a pragmatic effectiveness trial with a large sample. The rigorous pragmatic trial, with in-depth mixed methods, will demonstrate whether MT4C-In Care works across four Canadian provinces as well as the reasons and mechanisms underlying its effects. MT4C-In Care will be updated based on pragmatic trial results in Jan-Feb 2022.

Participants: Total of approximately 280 participants from four provinces will be recruited (100 each from Alberta and Ontario and 40 each from Saskatchewan and Manitoba). Each province will hire a recruitment specialist, and Alzheimer Societies and other community partners within each province will support recruitment of participants by including information in newsletters, distributing brochures, and/or attending support group meetings, etc. Recruited participants will be randomly assigned to the intervention and control group (140 participants each group) via a centralized web-based randomization service (REDCap).

Data Collection: Trained research assistants in each province will 1) track all participants' participation throughout the study, 2) conduct surveys with all participants by phone to assess whether or not the intervention was effective in improving outcomes over time, as compared to the control group, and 3) conduct in-depth telephone interview with five to fifteen participants (depending on the province; see below).

Number of Participants in Surveys and In-depth Interviews: Alberta and Ontario: surveys with all 100 participants and in-depth interviews with 15 participants; Saskatchewan and Manitoba: surveys with all 40 participants and in-depth interview with 5 participants.

Outcome Data Collection: Immediately before and after the intervention, outcome and process data will be collected from all caregivers.There will be 3 Data Collection Points: Baseline before the start of the intervention; 2-month follow up immediately post-intervention; 4 month follow up after the end of the intervention.

Data Analysis: Outcome will be analyzed (using Generalized Estimating Equations) to assess whether MT4C-In Care is effective in the intervention as compared to the control group over time. We anticipate that the intervention group will experience improved hope, mental health, quality of life, social support, and self-efficacy, and less loneliness and grief, as compared to the control group. 140 participants in each of the intervention and control groups will allow for rigorous testing of these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Family caregivers (≥18 years of age) of a person ≥65 years of age who has dementia that lives in a long-term care home
2. English-speaking
3. Has a valid email address and access to a computer and internet.

Exclusion Criteria:

1. Family caregivers of a person under the age of 65, who does not have dementia, or who does not reside in a long-term care home
2. Care partner has died
3. Non-English speaking
4. Under 18 years of age
5. No internet access or valid email

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the 12-item Short-Form Health Survey (SF-12v2) - Mental Component Summary Score at two and four months | Baseline, 2 months, 4 months
  The SF-12v2 is a measure of health related quality of life and provides 2 scores 1) Mental Component Summary Score (MCS) and 2) Physical Component Summary Score (PCS). MCS scores range from 0 to 100, higher scores indicate better mental health related quality of life

SECONDARY OUTCOMES:
Change from baseline in the 12-item Short-Form Health Survey (SF-12v2) - Physical Component Summary Score at 2 and 4 months. | Baseline, 2 months, 4 months
  The SF-12v2 is a measure of health related quality of life and provides 2 scores 1) Mental Component Summary Score (MCS) and 2) Physical Component Summary Score (PCS). PCS scores range from 0 to 100, higher scores indicate better physical health related quality of life
Change from baseline in the Herth Hope Index Score (HHI) at 2 and 4 months. | Baseline, 2 months, 4 months
  The HHI is a 12-item Likert-type scale used to measure hope. Items are scored from 1 "strongly disagree" to 4 "strongly agree", total scores range from 12 to 48 with a higher scores indicating greater hope. The items in the scale can be further divided into three factors of hope a) temporality and future, b) positive readiness and expectancy, and c) interconnectedness. Factor scores range from 4 to 16.
Change from baseline in the General Self-Efficacy Scale (GSES) at 2 and 4 months. | Baseline, 2 months, 4 months
  The GSES is a 10 item 4-point scale. The scale assesses a person's perceived self-efficacy-their belief that they can complete novel or difficult tasks or cope with diversity. Total scores range from 10 to 40 with higher scores indicating a greater level of self-efficacy.
Change from baseline in the Non Death Revised Grief Experience Inventory (NDRGEI) at 2 and 4 months. | Baseline, 2 months, 4 months
  The NDRGEI is a 22 item scale scored on a 6-point Likert scale from slightly disagree to strongly agree. The scale measures the grief experiences of persons anticipating a loss through four domains a) existential concerns (scores range 6-36), b) depression (scores range from 6-36), c) tension and guilt (scores range from 3-18), and d) physical distress (scores range from 7-42). The scale also offers a total grief score by calculating the sum of the four domains. The range for the total score is 22-132; higher scores indicate more grief.
Change from baseline in 3 item loneliness score at 2 and 4 months. | Baseline, 2 months, 4 months
  The Three-Item Loneliness Scale is an interviewer-administered questionnaire developed from the Revised University of California Los Angeles (UCLA) Loneliness Scale. Each question is rated on a 3-point scale: 1 = Hardly Ever; 2 = Some of the Time; 3 = Often. All items are summed to give a total score. Scores range from 3 to 9 (higher scores indicate more loneliness)
Change from baseline in Multidimensional Scale of Perceived Social Support at 2 and 4 months. | Baseline, 2 months, 4 months
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a brief research tool designed to measure perceptions of support from 3 sources: Family, Friends, and a Significant Other. The scale is comprised of a total of 12 items, with 4 items for each subscale. The total score is an average, calculated by summing all items (which could range from 12 to 84) and dividing by 12 (higher scores indicate more social support).

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Duggleby, PhD, Principal Investigator — University of Alberta; Hannah O'Rourke, PhD, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - University Of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duggleby W, Jovel Ruiz K, Ploeg J, McAiney C, Peacock S, Nekolaichuk C, Holroyd-Leduc J, Ghosh S, Brazil K, Swindle J, Forbes D, Woodhead Lyons S, Parmar J, Kaasalainen S, Cottrell L, Paragg J. Mixed-methods single-arm repeated measures study evaluating the feasibility of a web-based intervention to support family carers of persons with dementia in long-term care facilities. Pilot Feasibility Stud. 2018 Oct 31;4:165. doi: 10.1186/s40814-018-0356-7. eCollection 2018. PMID 30410783
- [Derived] Duggleby W, O'Rourke H, Swindle J, Peacock S, McAiney C, Baxter P, Thompson G, Dube V, Nekolaichuk C, Ghosh S, Holroyd-Leduc J. Study protocol: pragmatic randomized control trial of my tools 4 care- in care (MT4C-in care) a web-based tool for family Carers of persons with dementia residing in long term care. BMC Geriatr. 2020 Aug 10;20(1):285. doi: 10.1186/s12877-020-01690-w. PMID 32778059